CLINICAL TRIAL: NCT05203328
Title: Prospective Study to Evaluate High Flow Nasal Cannula With Monitored Anesthesia Care
Brief Title: Prospective Study to Evaluate High Flow Nasal Cannula With Monitored Anesthesia Care During EBUS Bronchoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-095
Record Dates: First submitted 2021-11-29; First posted 2022-01-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: EBUS; bronchoscopy; Vapotherm; high-flow nasal cannula; monitored anesthesia care (MAC)
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High flow nasal cannula oxygen (Experimental): High flow nasal cannula oxygen will be provided during the procedure using a Vapotherm device
  Interventions: Device: Vapotherm
- Regular nasal cannula (Active Comparator): Regular nasal cannula oxygen will be provided during the procedure
  Interventions: Device: Regular nasal canula

INTERVENTIONS:
Device: Vapotherm — Monitored anesthesia care with oxygen supplementation through a high-flow nasal cannula
  Other Names: High flow nasal cannula
  Arms: High flow nasal cannula oxygen
Device: Regular nasal canula — Monitored anesthesia care with oxygen supplementation through a regular nasal cannula
  Arms: Regular nasal cannula

SUMMARY:
Our objective is to assess whether the use of high flow nasal cannula (Vapotherm, Exeter, NH) with monitored anesthesia care (MAC) during an endobronchial ultrasound (EBUS) bronchoscopy procedure will lead to less procedure interruptions, less hypoxic episodes, shorter duration of hypoxic episodes and shorter procedural durations when compared to regular MAC using a regular nasal canula.

DETAILED DESCRIPTION:
Background:

MAC is a type of conscious sedation delivered by an anesthesiologist, during which different sedative medications are given, usually via the intravenous route, to obtain varying levels of sedation depending on the surgery or procedure. This is routinely done for all EBUS procedures at Cooper University Hospital. Since a MAC anesthesia does not include having a secure airway, occasionally the patient may develop episodes in which their oxygen level drops. During these episodes, the anesthesiologist will stop the procedure temporarily until the oxygen level returns to a normal range.

Often, changes in sedation amount is also required during this time. In a traditional MAC, the patient receives oxygen via a nasal cannula or a capnomask. If oxygen is delivered via a capnomask, the routine is to create a hole with scissors in the side of the capnomask in order to allow the bronchoscope into the patient's mouth. The Vapotherm is a breathing system used to deliver oxygen and remove carbon dioxide during anesthesia. The Vapotherm is a high flow nasal cannula that works by constantly providing humidified and heated high flow oxygen thereby creating positive end expiratory pressure that is useful for alveolar recruitment. It looks similar to nasal cannula but a little thicker and is also placed in the nostrils.

EBUS is a technique that uses ultrasound along with bronchoscopy to visualize the airway wall and structures adjacent to it. The clinical application and diagnostic benefits of EBUS have been well established, including diagnosis and staging of lung cancer. EBUS is usually performed under MAC for patient comfort.

The route of entry for the EBUS scope requires passage through the vocal cords and into the airways. The procedure tends to cause some discomfort and generally needs anesthesia to make people comfortable. Due to the amount of anesthesia required to subdue the airway reflexes for a smooth procedure, occasionally, the patient may become apneic or obstruct and not take adequate tidal volume breaths, leading to hypoxia. During these instances, the procedure is halted until the patient's oxygen levels return to baseline. We have noticed that anesthesiologists who prefer to use the Vapotherm in place tend to less often interrupt the procedure due to hypoxia.

Vapotherm high flow nasal cannula therapy is similar in efficacy to transtracheal catheters, which are intended to attenuate the effects of anatomical dead space on breathing efficiency. The mechanisms include washout of nasopharyngeal dead space, reduction of inspiratory resistance in the nasopharynx, improvement in airway and lung mechanics thereby providing methods to oxygenate without having to interrupt the procedure. All anesthesiologists at Cooper University Hospital are familiar with the Vapotherm high flow nasal cannula.

No research has been done in this field specifically regarding to EBUS. There is no anesthetic standard of care that is specific for an EBUS procedure. The anesthesia can be local anesthesia alone, with just topicalization of the airways, or MAC, or even general anesthesia with an endotracheal tube or a laryngeal mask airway. The choice is practitioner dependent.

Our experience has been that MAC with Vapotherm high flow leads to less procedural interruptions, less hypoxic episodes and shorter procedural durations.

Hypotheses:

Our hypothesis is that the use of the Vapotherm high flow nasal cannula with monitored anesthesia care (MAC) is associated with less procedure interruptions, less hypoxic episodes and shorter procedural durations.

Significance of the research:

If we can prove that the use of a Vapotherm high flow employed during MAC care leads to less procedure interruptions and shorter procedure durations, this would allow us to standardize the type of oxygen supply employed for EBUS in our institution and elsewhere. Less hypoxic episodes would benefit outcomes, lead to less recovery time and earlier discharges. Shorter procedural durations will create greater efficiency in the short procedure unit where the EBUS procedures are performed.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* patient undergoing EBUS bronchoscopy with moderate conscious sedation.

Exclusion Criteria:

* subjects with previous nasal surgeries
* subjects with oxygen saturation <90% on room air prior to procedure
* subjects who are pregnant
* subjects with known facial fractures or recent facial trauma
* subjects on any anticoagulation that cannot be discontinued prior to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of interruption during EBUS procedure for hypoxia | 1 day
  We will count the number of interruptions during EBUS procedure for hypoxia

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No